CLINICAL TRIAL: NCT05436561
Title: A Multiple-center Phase II Study to Evaluate the Clinical Outcome of Reduced Conditioning Regimen With Melphalan, Busulfan and Fludarabine for Patients >=55 Years With Myeloid Malignancies.
Brief Title: Reduced MBF Regimen for Patients >=55 Years With Myeloid Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBF-RIC-2022
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Disease-free Survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBF-RIC (Experimental): Patients with MBF-RIC as conditioning regimen
  Interventions: Drug: MBF-RIC

INTERVENTIONS:
Drug: MBF-RIC — Reduced intensity conditioning regimen with fludarabine, busulfan and melphalan
  Other Names: MBF100

SUMMARY:
In this multiple-center phase II study, the aim is to evaluate the clinical outcome of reduced intensity conditioning regimen with fludarabine (150mg/m2), busulfan (6.4mg/kg) and melphalan (100mg/m2) in patients with myeloid malignancies including AML, MDS and CMML >=55 years.

DETAILED DESCRIPTION:
Conditioning regimen with double alkylating agents such as busulfan + melphalan or Busulfan + thiotepa have been shown to improve the transplantation outcome in terms of lower relapse rate in various myeloid malignancies. In this multiple-center phase II study, the aim is to evaluate the clinical outcome of reduced intensity conditioning regimen with fludarabine (150mg/m2), busulfan (6.4mg/kg) and melphalan (100mg/m2) in patients with myeloid malignancies including AML, MDS and CMML >=55 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-65
* patients with HLA-matched sibling donors, 9-10/10 matched unrelated donors or haplo-identical donors.
* patients with AML in remission, or MDS in any stage, or CMML in any stage
* inform consent provided

Exclusion Criteria:

* patients with abnormal liver (>3N), renal (1.5N) or cardiac function
* patients with active infection

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 2 year
  survival without disease relapse or progression

SECONDARY OUTCOMES:
overall survival | 2 year
  survival
GVHD and relapse free survival | 2 year
  survival without graft failure, without relapse, without III-IV aGVHD and without mod/sev cGVHD.
Non-relapse mortality | 2 year
  Death without disease progression or relapse
Relapse | 2 year
  disease progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Hu, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, Shanghai Municipality
  - Shanghai No 6 Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No